CLINICAL TRIAL: NCT07160959
Title: Physical Exercise to Prevent Mild-cognitive Impairment Progression in Advanced Chronic Kidney Disease (CKD) and Dialysis Patients
Brief Title: Physical Exercise to Prevent Mild-cognitive Impairment in Patients With Kidney Disfunctions
Acronym: Exprecoimp-CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biogem s.c.ar.l. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ERA4HEALTHNUTRIBRAIN-086; ERA4HEALTH2024-NUTRIBRAIN (Other Grant/Funding Number: ERA4HEALTH Partnership)
Record Dates: First submitted 2025-08-16; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease (Stages 4 and 5); Mild Cognitive Impairment (MCI)
Keywords: Chronic Kidney Disease (CKD); stage G4-5 (CKD G4-5); dialysis; physical exercise; cognitive function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cognitive Dysfunction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Combined aerobic (walking) and resistance exercise group. Patients randomised to this group will receive a structured exercise program to be performed at least thrice a week for 26 weeks. The physical exercise intervention will be managed and supervised by the personnel of the centres participating in the trial. The training program will be personalised according to the patient's baseline functional capacity assessed by the 6-minute walking test (6MWT). The aerobic exercise will include seven bouts of 2-minute walking separated by 1-minute seated rest (up to 2-minute periods of resting in the Very Low category) at a slow to moderate speed. A smartphone application designed to guide the weekly increase in speed will also record the number of training sessions performed. An instructor will specifically instruct all patients to walk in rhythm with the metronome. The goal intensity for each session is 9-10 (light-fairly light) on the 20-point Borg RPE. The number of steps per session will
  Interventions: Behavioral: Exercise
- Placebo comparator (Placebo Comparator): The control group will undergo standard nephrology care that include optimization of medical therapy, nutritional advices, best dialysis practice.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Behavioral: Exercise — Patients will undergo a home-based low-intensity interval multi component exercise program including aerobic and strengthening exercise
  Arms: Experimental Arm
Other: Control (Standard treatment) — Patients will be treated with standard therapy based on their CKD stage
  Arms: Placebo comparator

SUMMARY:
This research project focuses on improving memory and thinking (cognitive function) in people with advanced chronic kidney disease (CKD), a condition that affects about 10% of adults and is often linked to cognitive problems. The study includes a clinical trial where patients will either receive standard care or follow a home-based exercise program involving walking and strength training, to see if regular physical activity can improve brain function. It also includes a large-scale analysis of data from the UK Biobank to explore blood and genetic markers, brain imaging, and lifestyle factors linked to cognitive health. The ultimate aim is to find effective, easy-to-implement strategies and early warning signs that could lead to better treatment and quality of life for people living with CKD.

DETAILED DESCRIPTION:
The project aims to test the impact of exercise programs on cognitive function in stage G 4-5 CKD and dialysis patients with MCI in a randomised clinical trial. A structured physical exercise program (walking exercise) effectively improved physical performance and quality of life in dialysis patients in a previous trial by us (see reference 6 by the investigators of this proposal). We will combine resistance and walking exercise in the active arm of the trial. In parallel with this trial, the project aims to test the cross-sectional and longitudinal relationship between physical activity (PAA) and the genetic and circulatory biomarkers of cognitive function and brain MRI in CKD patients and individuals without CKD in the UK Biobank.

Randomised clinical trial This trial will test a structured combined physical exercise program based on home-based aerobic (walking) exercise and resistance exercise maintained for 26 weeks on cognitive function in predialysis patients with advanced CKD (stages 4-5) and dialysis patients with MCI compared to the usual care (control group). In the two study arms, nutritional guidelines by KDIGO will be implemented, and nutrient intake will be periodically assessed. For this purpose, an App for CKD patients, including dietary advice and registering nutrients, will be adapted to the languages of centres in participating countries. Furthermore, body composition will be assessed during the study visits using validated bio-impedance spectroscopy instruments. Two-thirds of enrolees will be predialysis CKD patients and one-third dialysis patients (haemodialysis or peritoneal dialysis patients). Partners or caregivers to assist patients in the trial's exercise arm are requested explicitly for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* CKD at KDOQI stage 4-5
* concomitant MCI (MOCA - MMSE (17 < MoCA < 26) or (16 < MMSE < 24)

Exclusion Criteria:

* Absolute contraindication to exercise training (e.g. unstable angina, major amputation, severe heart failure, etc.)
* Known life expectancy < 6-month
* Uncorrected anemia (Hb <9 g/dl)
* Non-provision of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | Baseline; End of program (6-month); Follow up (12-month; 24-month)
  Cognitive function using the Alzheimer Disease Assessment Scale Cognitive 11 (ADAS-Cog-11)

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | Baseline and 6 months
  Blood Oxygenation Level-Dependent (BOLD) Signal will be collected through functional MRI executed according to the published standards
6-minute walking test | Baseline; End of program (6-month); Follow up (12-month; 24-month)
  The patients will be instructed to walk back and forth on a 20-meter corridor aiming at covering as much distance as possible. The total distance covered (6MWD) will be measured in meters
Quality of life assessment | Baseline; end of the program (6-month); Follow up (12-month; 24-month)
  Quality of life will be assessed by the short-form 36 (SF-36) questionnaire This is a generic questionnaire that contains 36 questions referring to 8 specific domains related to patient health over the previous 4 weeks
Lower limbs strength assessment | Baseline; end of the program (6-month); Follow up (12-month; 24-month)
  Lower limbs strength assessed by the 5-time sit-to-stand test Patients will raise up from a standard height chair with their arms folded across the chest five times as quickly as possible. The total time elapsed for completing the five repetitions is recorded in seconds
Handgrip strength | Baseline; End of program (6-month); Follow up (12-month; 24-month)
  Handgrip strength will be measured by a standard dynamometer. Peak value in kg for both arms will be collected
Body mass index assessment | Baseline, end of the program (6-month); follow up (12-month; 24-month)
  Body mass index Body composition will be assessed with direct measures of height and weight. Body mass index will be calculated as the ratio between weight (in kg) and the squared height (in meters)
Safety and tolerability | End of treatment (6-month)
  Number of participants with treatment-related adverse events as assessed by the CTCAE version 4.0
Long-term survival rate assessment | Baseline, end of treatment (6-month); follow up (12-month); follow up (18-month); Follow up (24-month); Follow up (36-month)
  Long-term survival rate All-cause mortality of the enrolled patients will be checked from the regional's datasets. In case of positive findings, the days elapsed from enrollment to the event will be recorded for additional analyses, as well as the reasons and the diagnoses.
Long-term hospitalizations assessment | Baseline, end of treatment (6-month); follow up (12-month); follow up (18-month); Follow up (24-month); Follow up (36-month)
  Long-term hospitalizations All-cause hospitalization will be checked from the regional's datasets. In case of positive findings, the days elapsed from enrollment to the event will be recorded for additional analyses, as well as the reasons and the diagnoses.

CONTACTS AND LOCATIONS:
Locations (6):
- Assistance Publique - Hôpitaux de Paris (AP-HP), Division of Geriatry, Paris, France
- Biogem, Ariano Irpino, Italy
- Lithuanian University of Health Sciences, Kaunas, Lithuania
- University Medical Center Groningen, Department of Nephrology, Groningen, Netherlands
- Medical University of Warsaw, Department of Nephrology, Dialysis and Internal Medicine, Warsaw, Poland
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be shared with investigators who will make a request to the Principal investigator immediately after the publication of the main study results.
Time Frame: after the publication of the main study results
Access Criteria: Scientists will be able to access supporting in formation, they will access the study protocol and the results.